CLINICAL TRIAL: NCT00123981
Title: The Impact of Avoiding Cardiopulmonary By-pass During Coronary Artery Bypass Surgery for Ischemic Heart Disease in Elderly Patients: The Danish On-pump, Off-pump Randomization Study (DOORS)
Brief Title: The Danish On-pump, Off-pump Randomization Study (DOORS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kim Houlind (Other)
Responsible Party: Sponsor-Investigator, Kim Houlind, Senior consultant, Associate Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTS-0001
Record Dates: First submitted 2005-07-25; First posted 2005-07-26 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Ischemic Heart Disease
Keywords: Off-pump Coronary Artery By-pass Grafting; Randomization; stroke; myocardial infarction; mortality; graft patency; quality of life
MeSH Terms: conditions — Myocardial Ischemia; Stroke; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CCABG (Active Comparator): Coronary artery bypass surgery using cardiopulmonary bypass
  Interventions: Procedure: Off-Pump Coronary Artery Bypass Grafting
- OPCAB (Experimental): Coronary artery bypass surgery NOT using cardiopulmonary bypass
  Interventions: Procedure: Off-Pump Coronary Artery Bypass Grafting

INTERVENTIONS:
Procedure: Off-Pump Coronary Artery Bypass Grafting

SUMMARY:
Background: Coronary artery bypass grafting (CABG) can be performed either with or without the use of cardiopulmonary bypass (CPB) to obtain myocardial re-vascularisation. The investigators hypothesize that CABG without the use of CPB may reduce the risk of perioperative death, stroke, myocardial infarction and other serious complications.

The aim of the present study is to compare the incidence of complications and the clinical efficacy of CABG with and without the use of CPB in elderly patients.

DETAILED DESCRIPTION:
Conventional coronary artery bypass grafting (CCABG) using cardiopulmonary bypass has for decades been applied to obtain myocardial re-vascularisation and, hence, improved quality of life and survival. It does, however, bear a risk of death, stroke, myocardial infarction and other serious complications.

During recent years, an equivalent operation performed on the beating heart without cardiopulmonary bypass (off-pump coronary artery bypass grafting, OPCAB) has gained popularity helped by the advent of mechanical stabilization devices and improved surgical techniques. Observational studies suggest that this technique is associated with a lower incidence of stroke, per operative arrhythmias and even mortality than conventional CCABG. This is especially the case in elderly patients and patients with significant co-morbidity.

Only few randomised, controlled trials have been conducted and most of these included mainly or only low-risk, relatively young patients. These studies have documented the safety and efficacy of OPCAB compared with CCABG, but none of the trials has had the statistical strength to determine whether the rate of serious complications is lower after OPCAB operations. One recent study found graft patency to be significantly lower after OPCAB than after CCABG operations.

The investigators find that there is a need of a larger scale randomised trial to compare the results of CCABG and OPCAB operations, especially in elderly patients. This patient group is poorly represented in earlier randomised trials, whereas observational studies and theoretical considerations imply that they may benefit the most from avoiding cardiopulmonary bypass.

Aims: Primarily, to compare the incidence of death, stroke and myocardial infarction after CCABG and OPCAB procedures in a population of elderly patients. Furthermore, to compare quality of life and graft patency, and cost- effectiveness after CCABG and OPCAB.

ELIGIBILITY:
Inclusion Criteria:

* Age seventy years or above
* Admitted for first time coronary artery bypass operation

Exclusion Criteria:

* Given information cannot be understood
* Aortic crossclamping not safe due to calcification
* Preoperative cardiac conditions demanding cardiopulmonary bypass
* Re-do cardiac surgery
* Patients requiring operation within the same day after conference

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 900 (Actual)
Dates: Start 2005-01; Primary Completion 2008-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
A combined endpoint of death + stroke + myocardial infarction within 30 days from operation | 30 days

SECONDARY OUTCOMES:
A combined endpoint of death + stroke + myocardial infarction during follow-up | 3 years
Patency of bypass grafts assessed by coronary angiography 6 months after the operation | 6 months
Total mortality and cardiac mortality during follow-up | 3 years
Need of new intervention for cardiac angina during follow-up | 3 years
Quality of life assessed by MOS SF-36 and EuroQol questionnaires 6 months and 3 years after the operation | 6 months and 3 years
Total hospital costs and costs of public care provided 6 months and 3 years after the operation and difference in costs per quality adjusted life year | 6 months and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim C Houlind, MD, PhD, Principal Investigator — Aarhus University Hospital; Poul E Mortensen, MD, Study Chair — Odense University Hospital
Locations (1):
- Dept. of Cardiothoracic and Vascular Surgery, Skejby Sygehus, Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Background] Houlind KC, Kjeldsen BJ, Terp KA, Madsen SN, Schmidt TA, Holme SJ, Mortensen PE. [Coronary artery bypass surgery without the use of a heart-lunch machine]. Ugeskr Laeger. 2005 May 9;167(19):2037-41. No abstract available. Danish. PMID 15960455
- [Derived] Houlind K, Fenger-Gron M, Holme SJ, Kjeldsen BJ, Madsen SN, Rasmussen BS, Jepsen MH, Ravkilde J, Aaroe J, Hansen PR, Hansen HS, Mortensen PE; DOORS Study Group. Graft patency after off-pump coronary artery bypass surgery is inferior even with identical heparinization protocols: results from the Danish On-pump Versus Off-pump Randomization Study (DOORS). J Thorac Cardiovasc Surg. 2014 Nov;148(5):1812-1819.e2. doi: 10.1016/j.jtcvs.2014.02.024. Epub 2014 Feb 8. PMID 24613160
- [Derived] Houlind K, Kjeldsen BJ, Madsen SN, Rasmussen BS, Holme SJ, Nielsen PH, Mortensen PE; DOORS Study Group. On-pump versus off-pump coronary artery bypass surgery in elderly patients: results from the Danish on-pump versus off-pump randomization study. Circulation. 2012 May 22;125(20):2431-9. doi: 10.1161/CIRCULATIONAHA.111.052571. Epub 2012 Apr 20. PMID 22523305
- [Derived] Houlind K, Kjeldsen BJ, Madsen SN, Rasmussen BS, Holme SJ, Schmidt TA, Haahr PE, Mortensen PE; DOORS study group. The impact of avoiding cardiopulmonary by-pass during coronary artery bypass surgery in elderly patients: the Danish On-pump Off-pump Randomisation Study (DOORS). Trials. 2009 Jul 4;10:47. doi: 10.1186/1745-6215-10-47. PMID 19575814
- See also: home page of the Danish Heart Foundation — http://www.hjerteforeningen.dk